CLINICAL TRIAL: NCT06644443
Title: BCMA-GPRC5D CAR-T Therapy in Relapsed or Refractory Multiple Myeloma：A Prospective, Single-center, Single-arm Phase I/IIa Clinical Trial
Brief Title: BCMA-GPRC5D CAR-T Therapy in Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-ONCO-028
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma in Relapse
Keywords: Neoplasms by Histologic Type; Neoplasms; Hemostatic Disorders; Vascular Diseases; Cardiovascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases; Multiple Myeloma; Neoplasms, Plasma Cell
MeSH Terms: conditions — Neoplasms by Histologic Type; Neoplasms; Hemostatic Disorders; Vascular Diseases; Cardiovascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases; Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental：Treatment group (Experimental): patients treated with BCMA-GPRC5D CAR-T cells
  Interventions: Biological: BCMA-GPRC5D CAR-T cells

INTERVENTIONS:
Biological: BCMA-GPRC5D CAR-T cells — patient was subjected to 2-5×10^6 BCMA-GPRC5D CAR-T cells/kg

SUMMARY:
At present, MM is still an incurable disease in general, and the vast majority of patients will eventually face disease recurrence or progression. Although CAR-T therapy targeting BCMA has shown advantages in the efficacy and safety of MM, for MM patients with BCMA negative or BCMA low expression, they still relapse after receiving targeted BCMA CAR T-cell therapy, and there is a problem of target escape. The specific high expression of GPRC5D in multiple myeloma cells makes it possible to combine BCMA and GPRC5D in the treatment of MM. This study aims to investigate the safety and efficacy of BCMA-GPRC5D CAR-T therapy in the treatment of relapsed or refractory MM.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a hematological malignant tumor characterized by clonal proliferation of abnormal plasma cells in the bone marrow. The incidence of MM is mainly in the middle and old age, and the incidence of MM in China has increased in recent years. At present, MM is still an incurable disease in general, and the vast majority of patients will eventually face disease recurrence or progression. Recurrent or refractory MM is still a thorny problem in the treatment of MM, which is an important factor for the survival of patients.Although CAR-T therapy targeting BCMA has shown advantages in the efficacy and safety of MM, for MM patients with BCMA negative or BCMA low expression, they still relapse after receiving targeted BCMA CAR T-cell therapy, and there is a problem of target escape. The specific high expression of GPRC5D in multiple myeloma cells makes it possible to combine BCMA and GPRC5D in the treatment of MM. This study aims to investigate the safety and efficacy of BCMA-GPRC5D CAR-T therapy in the treatment of relapsed or refractory MM.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (≥ 18 years old, ≤ 75 years old), gender is not limited;
2. The subject voluntarily participates in the research and signs the "Informed Consent" by himself or his legal guardian;
3. Definitely diagnosed as relapsed or refractory multiple myeloma: use chemotherapy regimens containing bortezomib, or chemotherapy regimens containing lenalidomide, the treatment is ineffective, or the disease progresses within 60 days after the end of the last chemotherapy;
4. The patient has one or more measurable multiple myeloma lesions, which must include any of the following:1) Serum M protein is greater than or equal to 0.5g / dl (10g / l) 2) Urine M protein is greater than or equal to 200 mg / 24 h serum FLC ratio is abnormal 3) Serum free light chain (FLC) ≧5 mg / dL (50 mg /L) 4) Plasmacytoma that can be measured by physical examination or imaging examination 5) Myeloma cells in bone marrow ≧10% by flow cytometry or immunohistochemical examination
5. After flow cytometry or immunohistochemical examination, myeloma cells have positive BCMA and GPRC5D expression;
6. No salvage chemotherapy was used within 4 weeks before cell therapy;
7. No antibody drug therapy was used within 2 weeks before cell therapy;
8. The ECOG score is 0-2 points;
9. The subject has no contraindications to peripheral blood apheresis;
10. The expected survival period is ≧12 weeks;
11. Female subjects of childbearing age must have a negative urine pregnancy test within 7 days prior to cell therapy and not during the lactation period; female or male subjects of childbearing age must take effective contraceptive measures throughout the study

Exclusion Criteria:

1. Those who have a history of allergies to any of the ingredients in cell products;
2. The following conditions in laboratory tests: including but not limited to serum total bilirubin ≥ 1.5 mg/dl; serum ALT or AST greater than 2.5 times the upper limit of normal; blood creatinine ≥ 2.0 mg/dl; hemoglobin<80g/l; does not rely on GCSF or other growth factors, the absolute neutrophil count is less than 1000 / mm3; no blood transfusion is required, and the platelet count is less than 30,000 / mm3;
3. According to the New York Heart Association (NYHA) cardiac function classification standards, patients with grade III or IV cardiac insufficiency; or echocardiographic examination of left ventricular ejection fraction (LVEF) <50%;
4. Abnormal lung function, blood oxygen saturation in indoor air<92%;
5. Myocardial infarction, cardiovascular angioplasty or stenting, unstable angina, or other serious clinical heart diseases within 12 months before enrollment;
6. Hypertension is grade 3 and the blood pressure is not well controlled by medication;
7. Patients with prolonged QT interval on ECG, patients with severe heart disease such as severe arrhythmia in the past;
8. Previously suffering from head injury, disturbance of consciousness, epilepsy, more serious cerebral ischemia or cerebral hemorrhage disease;
9. Need to use any anticoagulant (except aspirin);
10. Patients who need urgent treatment due to tumor progression or spinal cord compression;
11. Patients with CNS metastasis or CNS involvement symptoms (including cranial neuropathy and extensive disease or spinal cord compression);
12. The investigator determines that there are serious complications or diseases that increase the risk of the subject or affect the research, including but not limited to, for example: liver cirrhosis, recent major trauma, etc.;
13. After allogeneic hematopoietic stem cell transplantation;
14. Plasma cell leukemia;
15. Before apheresis and within 2 weeks before CAR-T cell infusion, apply more than 5 mg/d of prednisone (or an equivalent amount of other corticosteroids);
16. Patients with autoimmune diseases, immunodeficiencies or other patients who need immunosuppressive therapy;
17. There is an uncontrolled active infection;
18. Live vaccination within 4 weeks before enrollment;
19. HIV, HBV, HCV and TPPA/RPR infected persons, and HBV carriers;
20. The subject has a history of alcoholism, drug abuse or mental illness;
21. The subject has participated in any other clinical research within 3 months before joining this clinical research;
22. The researcher believes that the subjects have other conditions that are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-07-14 (Estimated); Study Completion 2026-07-14 (Estimated)

PRIMARY OUTCOMES:
TEAEs | From date of initial treatment to the 30 days after treatment
  Adverse events during treatment

SECONDARY OUTCOMES:
Disease-related clinical responses | From data of enrollment until the data of clinical responses,up to 2 years.
  Disease-related clinical responses include sCR/CR/VGPR/PR/MR/SD/PD

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Guo, Doctor, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Shenzhen University General Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No